CLINICAL TRIAL: NCT03946111
Title: Cognitive-Behavioral and Pharmacologic Treatment of Binge-Eating Disorder and Obesity
Brief Title: Cognitive-Behavioral and Pharmacologic (LDX) Treatment of Binge-Eating Disorder and Obesity: Medication Change for Non-Responders
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000022480_a; 1R01DK114075-01A1 (NIH)
Record Dates: First submitted 2019-04-22; First posted 2019-05-10 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Binge-Eating Disorder; Obesity
MeSH Terms: conditions — Binge-Eating Disorder; Obesity | interventions — bupropion hydrochloride, naltrexone hydrochoride drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Naltrexone/Bupropion (Experimental)
  Interventions: Drug: Naltrexone and Bupropion
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Naltrexone and Bupropion — Participants randomly assigned to this arm will receive 12 weeks of Naltrexone and Bupropion medication.
  Arms: Naltrexone/Bupropion
Other: Placebo — Participants randomly assigned to this arm will receive 12 weeks of an inactive placebo.
  Arms: Placebo

SUMMARY:
This study will test the relative efficacy and effectiveness of the combination of naltrexone and bupropion (NB) medication as a treatment for binge-eating disorder (BED) in patients with obesity. This is a controlled test of whether, amongst non-responders to acute treatments, NB medication results in superior outcomes compared with placebo.

DETAILED DESCRIPTION:
Obesity is a heterogeneous problem and research has highlighted the particular significance of a subgroup with binge-eating disorder (BED), the most prevalent formal eating disorder. Improved treatments for patients with obesity and BED are needed that can produce sustained clinical outcomes and promote weight loss. This study RCT will provide new and novel findings from a controlled test, amongst non-responders to acute treatments, whether Naltrexone/Bupropion medication results in superior and longer-term outcomes than placebo.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 64 years old
* Meets DSM-5 criteria for binge-eating disorder
* BMI 27-30 with a controlled obesity-related co-morbidity; or BMI ≥ 30 and <50
* Medically cleared as determined by EKG and medical record review
* Available for the duration of the treatment and follow-up (18 months)
* Read, comprehend, and write English at a sufficient level to complete study-related materials
* Able to travel to study location (New Haven, CT) for weekly visits

Exclusion Criteria:

* Previous history of problems with LDX or other stimulants
* Current psychostimulant use or use of any medication for ADHD
* Current use of study medications: LDX (Vyvanse), Bupropion (Wellbutrin, Zyban), Naltrexone, or Contrave
* History of congenital heart disease, known structural cardiac abnormalities, cardiomyopathy, serious heart arrhythmia, coronary artery disease, cerebrovascular pathology including stroke, exertional chest pain, uncontrolled high blood pressure, and other serious heart problems.
* History of severe renal, hepatic, neurological, or chronic pulmonary disease or other serious, unstable medical disorder.
* Current uncontrolled hypertension
* Current uncontrolled type I or II diabetes mellitus
* Current uncontrolled thyroid illness
* Gallbladder disease
* Co-occurring severe mental illness requiring hospitalization or intensive treatment
* Endorses current active suicidal or homicidal ideation with intent or plan
* History or current alcohol or substance use disorder (smoking is not exclusionary)
* Predisposition to seizures
* History of anorexia nervosa or bulimia nervosa, or currently regularly self-inducing vomiting
* Currently taking MAOI, SSRI or strong inhibitors of CYP2D6
* History of allergy or sensitivity to the study medication or stimulant medications
* Current use of medications contraindicated with the study medications
* Currently breast feeding or pregnant, or not willing to use reliable form of contraception
* Currently taking opioid pain medications or drugs
* Currently using effective treatment (evidence-based therapeutic or psychopharmacologic) for eating and/or weight loss
* Currently participating in another clinical study in which the participant is or will be exposed to an investigational or a non-investigational drug or device
* Medical status judged by study physician as contraindication

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Grilo, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale Department of Psychiatry, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naltrexone/Bupropion | Placebo
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone/Bupropion | Placebo | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (0.0) | 43 (19.8) | 44.33 (14.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Binge-Eating Frequency
Description: Binge-eating frequency is a continuous variable of binge-eating episodes assessed using interview (Eating Disorder Examination interview). The Eating Disorder Examination uses a 28 day recall of eating behavior. The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM -5) defines binge-eating as "eating, in a discrete period of time an amount of food that is definitely larger than most people would eat during a similar period of time and under similar circumstances and a sense of loss of control over eating during the episode." The number of episodes that meet this description will be counted and totaled.
Time Frame: From baseline interview at study enrollment to 3 months after the 12-week treatment.
Measure: Mean (Standard Deviation); unit: episodes per past 28 days
Arm/Group | Naltrexone/Bupropion | Placebo
Number analyzed (Participants) | 1 | 2
episodes per past 28 days | -14 (0) | -17.00 (18.38)

2. Primary Outcome: Change in Binge-Eating Frequency
Description: as for outcome 1
Time Frame: From post-treatment to the 6-month follow-up
Measure: Mean (Standard Deviation); unit: episodes per past 28 days
Arm/Group | Naltrexone/Bupropion | Placebo
Number analyzed (Participants) | 1 | 2
episodes per past 28 days | 0 (0) | 3 (0)

3. Primary Outcome: Change in Binge-Eating Frequency
Description: as for outcome 1
Time Frame: From post-treatment to the 12-month follow-up
Measure: Mean (Standard Deviation); unit: episodes per past 28 days
Arm/Group | Naltrexone/Bupropion | Placebo
Number analyzed (Participants) | 1 | 2
episodes per past 28 days | 4 (0) | 1.50 (2.12)

4. Primary Outcome: Percent Change in Weight
Description: Negative values indicate weight loss and positive values indicate weight gain.
Time Frame: From baseline interview at study enrollment to 3 months after the 12-week treatment.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Naltrexone/Bupropion | Placebo
Number analyzed (Participants) | 1 | 2
percent change | 2.71 (0) | -1.73 (11.35)

5. Primary Outcome: Percent Change in Weight
Description: Negative values indicate weight loss and positive values indicate weight gain.
Time Frame: From post-treatment to the 6-month follow-up
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Naltrexone/Bupropion | Placebo
Number analyzed (Participants) | 1 | 2
percent change | 5.82 (0.0) | 5.61 (8.88)

6. Primary Outcome: Percent Change in Weight
Description: Negative values indicate weight loss and positive values indicate weight gain.
Time Frame: From post-treatment to the 12-month follow-up
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Naltrexone/Bupropion | Placebo
Number analyzed (Participants) | 1 | 2
percent change | 12.33 (0.0) | 3.32 (5.24)

7. Secondary Outcome: Binge-Eating Remission
Description: Categorical: zero binges/28 days
Time Frame: 12-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Naltrexone/Bupropion | Placebo
Number analyzed (Participants) | 1 | 2
Participants | 1 | 2

8. Secondary Outcome: Binge-Eating Remission
Description: Categorical: zero binges/28 days
Time Frame: 6-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Naltrexone/Bupropion | Placebo
Number analyzed (Participants) | 1 | 2
Participants | 1 | 0

9. Secondary Outcome: Binge-Eating Remission
Description: Categorical: zero binges/28 days
Time Frame: 12-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Naltrexone/Bupropion | Placebo
Number analyzed (Participants) | 1 | 2
Participants | 0 | 1

10. Secondary Outcome: Change in Eating-Disorder Psychopathology (Continuous)
Description: Eating-disorder psychopathology is assessed by the global score of the Eating Disorder Examination/Eating Disorder Examination-Questionnaire. Scores range from 0-6 (0=no eating-disorder psychopathology; 6=severe eating-disorder psychopathology).
Time Frame: From baseline interview at study enrollment to 3 months after the 12-week treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone/Bupropion | Placebo
Number analyzed (Participants) | 1 | 2
score on a scale | -1.07 (0.0) | -0.33 (2.49)

11. Secondary Outcome: Change in Eating-Disorder Psychopathology (Continuous)
Description: Eating-disorder psychopathology is a continuous variable as assessed by the global score of the Eating Disorder Examination/Eating Disorder Examination-Questionnaire. Scores range from 0-6 (0=no eating-disorder psychopathology; 6=severe eating-disorder psychopathology).
Time Frame: From post-treatment to the 6-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone/Bupropion | Placebo
Number analyzed (Participants) | 1 | 2
score on a scale | 0.14 (0.0) | 0.09 (0.36)

12. Secondary Outcome: Change in Eating-Disorder Psychopathology (Continuous)
Description: as for outcome 11
Time Frame: From post-treatment to the 12-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone/Bupropion | Placebo
Number analyzed (Participants) | 1 | 2
score on a scale | 0.76 (0) | -0.22 (0.69)

13. Secondary Outcome: Change in Depressive Symptoms
Description: Depressive symptoms is a continuous variable of depressive symptomatology as assessed by the self-report measure, the Beck Depression Inventory - Second Edition. Scores range from 0-63 (0=no depressive symptoms, 63=greater depressive symptoms).
Time Frame: From baseline interview at study enrollment to 3 months after the 12-week treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone/Bupropion | Placebo
Number analyzed (Participants) | 1 | 2
score on a scale | -1.0 (0.0) | -5.50 (4.95)

14. Secondary Outcome: Change in Depressive Symptoms
Description: as for outcome 13
Time Frame: From post-treatment to the 6-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone/Bupropion | Placebo
Number analyzed (Participants) | 1 | 2
score on a scale | -7.0 (0.0) | -2.50 (2.12)

15. Secondary Outcome: Change in Depressive Symptoms
Description: as for outcome 13
Time Frame: From post-treatment to the 12-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone/Bupropion | Placebo
Number analyzed (Participants) | 1 | 2
score on a scale | -1.0 (0.0) | 2.50 (2.12)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Naltrexone/Bupropion | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naltrexone/Bupropion (N=1) | Placebo (N=2)
Constipation (Gastrointestinal disorders) | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0
Dizziness (General disorders) | 0 | 0
Headache (General disorders) | 0 | 0
Insomnia (General disorders) | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT03946111/Prot_SAP_002.pdf
  • Informed Consent Form (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT03946111/ICF_001.pdf